CLINICAL TRIAL: NCT02859259
Title: Relative Bioavailability Study of BMS-626529 Administered as Prodrug BMS-663068 From 150-mg Low-dose Extended-release Tablets Compared to 600-mg Reference Extended-release Tablet in Healthy Subjects
Brief Title: A Study of the Relative Bioavailability of BMS-626529 Administered as BMS-663068 From 150mg Low-dose Extended-release Tablets Compared to 600mg Reference Extended-release Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 206219; AI438-080 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2016-07-28; First posted 2016-08-09 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — fostemsavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A: reference extended-release (ER) 1 tablet at 600mg (Experimental): A single dose of BMS-663068 administered orally as specified
  Interventions: Drug: BMS-663068 (1 tablet at 600 mg)
- Treatment B: low-dose ER 4 tablets at 150mg (Experimental): A single dose (4 tablets) of BMS-663068 administered orally as specified
  Interventions: Drug: BMS-663068 (4 tablets at 150 mg each tablet)

INTERVENTIONS:
Drug: BMS-663068 (1 tablet at 600 mg) — BMS-663068 (1 tablet at 600 mg). A single dose of BMS-663068 administered orally as specified.
  Arms: Treatment A: reference extended-release (ER) 1 tablet at 600mg
Drug: BMS-663068 (4 tablets at 150 mg each tablet) — BMS-663068 (4 tablets at 150 mg each tablet). A single dose (4 tablets) of BMS-663068 administered orally as specified.
  Arms: Treatment B: low-dose ER 4 tablets at 150mg

SUMMARY:
An oral dose in healthy subjects to determine the relative bioavailabilty of BMS-626529 administered as BMS-663068

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Target Population: Healthy subjects as determined by no clinically significant deviation from normal in medical and surgical history, physical examination, vital sign measurements, 12-lead ECG measurements and clinical laboratory test results. Body mass index (BMI) of 18.0 to 32.0 kg/m².
3. Subject Re-enrollment: This study permits the re-enrollment of a subject that has discontinued the study as a pre-treatment failure (i.e., subject has not been randomized/ has not been treated). If re-enrolled, the subject must be re-consented.
4. Age: Males and Females, ages 18 or age of majority to 50 years, inclusive.
5. Reproductive Status: Women of childbearing potential (WOCBP) must have a negative serum/urine (urine test not allowed at screening and Day -1 of Period 1) pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours prior to the start of study drug. Women must not be breastfeeding. Women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug (60 hours) plus 30 days (duration of ovulatory cycle) for a total of 33 days post-treatment completion. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of study drug (60 hours). In addition, male subjects must be willing to refrain from sperm donation during this time. Azoospermic males are exempt from contraceptive requirements. Women of childbearing potential who are continuously not heterosexually active are also exempt from contraceptive requirements, and still undergo pregnancy testing as described in this section.

Exclusion Criteria:

1. Medical History and Concurrent Diseases: History of any chronic or acute illness, gastrointestinal disease, gastrointestinal surgery within less than 4 weeks of dosing, blood donation within 4 weeks of dosing, blood transfusion within 4 weeks of dosing, smoking within less than 12 months prior to dosing, alcohol abuse, inability to tolerate oral medication, or inability to be venipunctured. Any other sound medical, psychiatric and/or social reason as determined by the investigator.
2. Physical and Laboratory Test Findings: Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs measurements, ECGs, or clinical laboratory determinations beyond what is consistent with the target population.
3. Exposure to any investigational drug or placebo within 4 weeks of study drug administration.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-08-12 (Actual); Primary Completion 2016-08-12 (Actual); Study Completion 2016-08-12 (Actual)

PRIMARY OUTCOMES:
Bioavailability of BMS-626529 from low-dose ER tablet formulation of BMS-663068 relative to the reference ER tablet formulation. | Approximately 8 days

SECONDARY OUTCOMES:
Safety and Tolerability as assessed by the Incidence of Serious Adverse Events (SAEs), Adverse Events (AEs), AEs leading to discontinuation, and the results of electrocardiogram tests (ECGs), vital signs, physical exams, and clinical laboratory tests. | Approximately 8 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No